CLINICAL TRIAL: NCT03917524
Title: The Feasibility of Circulating Tumor Cells Isolation for Transcriptomes and Genome-wide Associated Analysis in Post-surgically High-risk Oral Cavity Cancer Patients and Its Clinical Significance.
Brief Title: Feasibility of CTCs Isolation for Transcriptomes and Genome Wide Associated Analysis in Post-OP High Risk OSCC Patients.
Acronym: CTC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: CTCNGS002; MOST104-2314-B-182A-073-MY3 (Other: Grantor or Funder MOST104-2314-B-182A-073-MY3)
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Oral Cavity Squamous Cell Carcinoma
Keywords: Oral Cavity Cancer; Circulating Tumor Cells; Whole-genome analysis; transcriptomes; distant metastasis; locoregional recurrence; second primary tumor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- no need for any adjuvant therapy: Patients with oral cavity squamous cell carcinoma post-surgery no need for any adjuvant therapy
- with risk factors: Patients with oral cavity squamous cell carcinoma post-surgery with major risk factor(s) or 2 minor risk factors Stratification by Risk factors, alcohol, betel nut chewing and cigarette use status

SUMMARY:
Anti-cancer treatments have been thought to be closely related to their unique genetic alterations. In the past few years, the investigator have used cDNA microarray to delineate the transcriptome profiles of differentially-expressed genes between OSCC tumors and normal epithelium. By supervised hierarachical clustering analysis, the investigator further analyzed and validated the differentially-expressed genes for OSCC tumors. In the investigators' previous research, the investigators have used this strategy to analyze the potential tissue proteins associated with OSCC tumors, indicating the feasibility of this strategy. However, gene detection is a great limitation and challenge in CTCs researches owing to the small number of isolated cells by traditional methods. Fortunately, by means of the investigators' developing high-purity CTCs isolation techniques, some preliminary data implied that isolated CTCs by this method could achieve the criteria of Whole-genome analysis (WGA), which brings the investigators' passion for further investigation.

DETAILED DESCRIPTION:
First Year

1. Negative Selection Method 2. Positive Selection method (Dynabeads) 3. ODEP devices 4. Flow Cytometry and Sorting System 5. Cell lines for Positive control Second Year &Third year

1. Clinical Trial, Patient Enrollment and Design of Schedule

   The Inclusion criteria and aims are as followings:
   1. Patients with oral cavity squamous cell carcinoma (n=180), with age at diagnosis ≥ 20 years, will be enrolled before surgery at Ear-Nose-Throat department inpatient or outpatient service by Dr. Liao, Dr. Hsieh, Dr. Wang and co-PIs.
   2. All patients will be subgrouped by pathologic features and risk factors Group A (n=90): OSCC, post-surgery, no need for any adjuvant therapy Group B (n=90): OSCC, post-surgery, with major risk factor(s) or 2 minor risk factors Stratification by Risk factors, alcohol, betel nut chewing and cigarette use status
   3. Testing: Circulating tumor cells (CTCs) (x4) and NGS for WGA and transcriptomes (x4)
   4. Endpoints: Loco-regional recurrence, one-year distant metastasis rate, death, second primary tumor occurrence.
   5. Exclusion criteria are: (1) Patient's refusal; (2) Poor compliance, cannot cooperate for blood sampling for CTCs isolation as time schedule or clinical treatment or follow-up (3) Difficult blood sampling; (4) No more needs for CTCs evaluation, decided by clinicians.
2. Whole-Genome Analysis for Cancer Tissue Samples/Circulating Tumor Cells When needed, OncoScan™ FFPE Express Extraction will be performed

   Requirements need to be observed when submitting FFPE slices:

   Slices should be sent in 1.5mL conical vials Tumor samples in sections should have a surface area of 100 square mm (Minimum) to 1000 square mm (Maximum).

   Normal samples in sections should have a surface area of 200 square mm (Minimum) to 1000 square mm (Maximum).

   Section thickness should be 10 micron. The range of sections acceptable per sample is 2-6. Slices for OncoScan analysis and immunohistochemistry study are separated; and will be doubly charged by the Dep. of Clinical Pathology.

   The QIAamp DNA FFPE Tissue Kit is optimized for purification of DNA from FFPE tissue sections.

   OncoScan™ Express Samples will be performed in Chang Gung Memorial Hospital 1J GMRCL CoreLab or Chang Gung University Labs for whole-genome analysis.
3. Negative Selection Method
4. Positive Selection method (Dynabeads)
5. ODEP devices
6. Flow Cytometry and Sorting System

ELIGIBILITY:
Inclusion Criteria:

* Patients with oral cavity squamous cell carcinoma (n=180), with age at diagnosis ≥ 20 years, will be enrolled before surgery at Ear-Nose-Throat department inpatient or outpatient service by Dr. Liao, Dr. Hsieh, Dr. Wang and co-PIs.

Exclusion Criteria:

* (1) Patient's refusal; (2) Poor compliance, cannot cooperate for blood sampling for CTCs isolation as time schedule or clinical treatment or follow-up (3) Difficult blood sampling; (4) No more needs for CTCs evaluation, decided by clinicians.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with oral cavity squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | one year
  Measure response or progression events via all available imaging studies, including Chest-Xray, CT scans, or MRI, Positron Emission Tomography(PET)study. The relationship between CTCs number and time from CTCs checkpoint to disease progression will be analyzed.

SECONDARY OUTCOMES:
Overall survival | one year
  All causes of death would be documented and the relationship between CTCs number and time from CTCs checkpoint to death will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ta Liao, MD, Principal Investigator — Division of Otolaryngology, Chang Gung Memorial Hospital at Linkou
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan